CLINICAL TRIAL: NCT01136382
Title: Phase 2, Double-blind, Randomized, Parallel-group, Placebo-controlled, Multicenter Study, Comparing Budesonide pMDI 160 ug Bid With Placebo: a 6-week Efficacy and Safety Study in Children Aged 6 to <12 Years With Asthma
Brief Title: A 6-week Study in Asthmatic Children Aged 6 to <12 Yrs Comparing Budesonide pMDI 160ug Twice Daily With Placebo
Acronym: CHASE 1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D589GC00001
Record Dates: First submitted 2010-06-01; First posted 2010-06-03 (Estimated); Results first posted 2014-07-21 (Estimated); Last update posted 2014-08-01 (Estimated); Status verified 2014-07

CONDITIONS: Asthma
Keywords: asthma, children, budesonide pMDI
MeSH Terms: conditions — Asthma | interventions — Budesonide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Budesonide pMDI 160 ug bid (80 ug x 2 inhalations bid)
  Interventions: Drug: budesonide
- 2 (Placebo Comparator): Placebo pMDI 2 inhalations bid
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: budesonide — pMDI, inhalation, bid, 6 weeks
  Arms: 1
Drug: placebo — pMDI, inhalation, bid, 6 weeks
  Arms: 2

SUMMARY:
This purpose of the study is to investigate if budesonide pMDI 160 �g twice a day during 6 weeks is effective and safe in treating asthmatic children aged 6 to <12 years

DETAILED DESCRIPTION:
Phase 2, double-blind, randomized, parallel-group, placebo-controlled, multicenter study, comparing budesonide pMDI 160 �g bid with placebo: a 6-week efficacy and safety study in children aged 6 to <12 years with asthma

ELIGIBILITY:
Inclusion Criteria:

* Has a documented clinical diagnosis of asthma for at least 6 months prior to Visit 2 that has required daily inhaled corticosteroid in the low dose range OR LTRA as monotherapy for at least 30 days prior to Visit 2.
* Has a morning clinic pre-bronchodilator FEV1 measured at least 6 hours after the last dose of inhaled short acting beta agonist of greater than or equal to 70% and less than or equal to 95% of predicted normal
* Demonstrated reversibility of FEV1 of ≥12% from pre short acting beta agonist level within 15 to 30 minutes after administration of a standard dose of short acting beta agonist OR has a documented reversibility of ≥ 12 % within 12 months prior to Visit 2.

Exclusion Criteria:

* Has been hospitalized at least once or required emergency treatment (was seen in the emergency room or had an urgent care visit) more than once for an asthma-related condition during the 6 months prior to Visit 2
* Has required treatment with systemic corticosteroids (eg, oral, parenteral, or rectal) for any reason within the 12 weeks prior to Visit 2

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 304 (Actual)
Dates: Start 2010-07; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Göran Eckerwall, MD, Study Director — AZ R&D Mölndal
Locations (87):
- United States (57):
  - Research Site, Scottsdale, Arizona
  - Research Site, Fresno, California
  - Research Site, Granada Hills, California
  - Research Site, Huntington Beach, California
  - Research Site, Mission Viejo, California
  - Research Site, Orange, California
  - Research Site, Palmdal, California
  - Research Site, Rolling Hills Estate, California
  - Research Site, San Diego, California
  - Research Site, Stockton, California
  - Research Site, Centennial, Colorado
  - Research Site, Colorado Springs, Colorado
  - Research Site, Denver, Colorado
  - Research Site, Coral Gables, Florida
  - Research Site, Orange City, Florida
  - Research Site, Sarasota, Florida
  - Research Site, Albany, Georgia
  - Research Site, Gainesville, Georgia
  - Research Site, Normal, Illinois
  - Research Site, Overland Park, Kansas
  - Research Site, Bethesda, Maryland
  - Research Site, North Dartmouth, Massachusetts
  - Research Site, Ypsilanti, Michigan
  - Research Site, Plymouth, Minnesota
  - Research Site, Columbia, Missouri
  - Research Site, St Louis, Missouri
  - Research Site, Bozeman, Montana
  - Research Site, Bellevue, Nebraska
  - Research Site, Omaha, Nebraska
  - Research Site, Ocean City, New Jersey
  - Research Site, Skillman, New Jersey
  - Research Site, Teaneck, New Jersey
  - Research Site, Rockville Centre, New York
  - Research Site, High Point, North Carolina
  - Research Site, Canton, Ohio
  - Research Site, Cincinnati, Ohio
  - Research Site, Cleveland, Ohio
  - Research Site, Sylvania, Ohio
  - Research Site, Toledo, Ohio
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Gresham, Oregon
  - Research Site, Lake Oswego, Oregon
  - Research Site, Medford, Oregon
  - Research Site, Portland, Oregon
  - Research Site, Altoona, Pennsylvania
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Upland, Pennsylvania
  - Research Site, Charleston, South Carolina
  - Research Site, Dallas, Texas
  - Research Site, El Paso, Texas
  - Research Site, Fort Worth, Texas
  - Research Site, Georgetown, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Waco, Texas
  - Research Site, Richmond, Virginia
  - Research Site, Greenfield, Wisconsin
  - Research Site, West Allis, Wisconsin
- Bulgaria (3):
  - Research Site, Plovdiv
  - Research Site, Rousse
  - Research Site, Sofia
- Hungary (12):
  - Research Site, Budapest
  - Research Site, Debrecen
  - Research Site, Győr
  - Research Site, Kiskunhalas
  - Research Site, Marcali
  - Research Site, Miskolc
  - Research Site, Nyíregyháza
  - Research Site, Sopron
  - Research Site, Szeged
  - Research Site, Szigetvár
  - Research Site, Törökbálint
  - Research Site, Zalaegerszeg
- Latvia (3):
  - Research Site, Ogre
  - Research Site, Rēzekne
  - Research Site, Riga
- Poland (5):
  - Research Site, Bialystok
  - Research Site, Częstochowa
  - Research Site, Karpacz
  - Research Site, Lodz
  - Research Site, Pabianice
- Slovakia (2):
  - Research Site, Bratislava
  - Research Site, Lučenec
- South Africa (5):
  - Research Site, Krugersdorp, Gauteng
  - Research Site, Durban, KwaZulu-Natal
  - Research Site, Pietermariztburg, KwaZulu-Natal
  - Research Site, Claremont, W Cape
  - Research Site, Panorama, W Cape

REFERENCES:
- [Derived] Meltzer EO, Pearlman DS, Eckerwall G, Uryniak T, DePietro M, Lampl K. Efficacy and safety of budesonide administered by pressurized metered-dose inhaler in children with asthma. Ann Allergy Asthma Immunol. 2015 Dec;115(6):516-22. doi: 10.1016/j.anai.2015.09.007. Epub 2015 Oct 13. PMID 26460293

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This multicenter study was conducted in Bulgaria, Hungary, Latvia, Poland, Slovakia, South Africa, and the United States between 07 August 2011 and 05 April 2013.
Pre-assignment Details: The study consisted of a screening visit (Visit 1), an enrollment visit (Visit 2), a 7- to 21-day run-in/qualification period, a randomization visit (Visit 3), and 6 further weekly visits during a treatment period of 6 weeks. A telephone follow-up was conducted approximately 2 weeks after the final study visit.
Groups:
- Placebo: Placebo pMDI bid
- Budesonide: Budesonide pMDI 160 mcg bid
Period: Overall Study
Arm/Group | Placebo | Budesonide
Started | 152 | 152
Completed | 92 | 121
Not Completed | 60 | 31
Not completed — Other | 8 | 3
Not completed — Study-Specific Withdrawal Criteria | 48 | 25
Not completed — Severe Non-Compliance to Protocol | 0 | 2
Not completed — Withdrawal by Subject | 4 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Budesonide | Total
Number analyzed (Participants) | 152 | 152 | 304
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.0 (1.62) | 9.0 (1.63) | 9.0 (1.62)
Age, Customized [Number; unit: participants]
  6 to <8 years | 33 | 33 | 66
  8 to- <12 years | 119 | 119 | 238
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 58 | 54 | 112
  Male | 94 | 98 | 192
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino | 10 | 11 | 21
  Native Hawaiian/Pacific Islander | 1 | 0 | 1
  African American | 7 | 9 | 16
  Asian (other than Chinese and Japanese) | 0 | 2 | 2
  Not Applicable | 128 | 126 | 254
  Other | 6 | 4 | 10
Forced expiratory volume in 1 second (FEV1) [Mean (Standard Deviation); unit: liters] | 1.70 (0.416) | 1.69 (0.388) | 1.70 (0.401)

OUTCOME MEASURES:

1. Primary Outcome: Change in Morning Peak Expiratory Flow (PEF) From Baseline to the Treatment Period Average
Description: The peak expiratory flow rate is the maximal rate that a person can exhale during a short maximal expiratory effort after a full inspiration. Baseline was calculated using the mean of the data recorded during the last 7 days of the run-in period, and the treatment period average was calculated as the mean of all available data recorded during the entire treatment period.
Time Frame: Baseline to 6 weeks
Population: The efficacy analysis set consisted of all patients who were randomized, received at least 1 dose of study medication, and contributed data for at least 1 efficacy endpoint.
Measure: Least Squares Mean (Standard Error); unit: liters/minute
Arm/Group | Placebo | Budesonide
Number analyzed (Participants) | 151 | 151
liters/minute | 4.1 (3.19) | 17.8 (3.24)
Statistical Analysis 1: Comparison: Placebo vs Budesonide; Change from baseline to treatment period average was analyzed using an analysis of covariance (ANCOVA) model with terms for treatment, age group (<8 years and ≥8 years of age) and country with baseline as a covariate; Test type: Superiority or Other; p < 0.0001, ANCOVA — To address multiplicity, a step-down procedure was used. If the treatment difference for the primary variable, morning PEF, was statistically significant (p<0.05), then the key secondary variable, FEV1, was tested at the 0.05 level of significance; LS mean difference = 13.6, 95% CI 2-sided [7.5 to 19.7], Standard Error of Mean 3.10

2. Secondary Outcome: Change in Forced Expiratory Volume in 1 Second (FEV1) From Baseline to Treatment Period Average
Description: FEV1 is the volume exhaled during the first second of a forced expiratory maneuver started from the level of total lung capacity. Baseline was defined as the pre-dose assessment value measured at randomization (Visit 3), and the treatment period average was calculated as the mean of all available data recorded during the entire treatment period.
Time Frame: Baseline to 6 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | Placebo | Budesonide
Number analyzed (Participants) | 149 | 152
liters | 0.00 (0.023) | 0.06 (0.023)
Statistical Analysis 1: Comparison: Placebo vs Budesonide; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0047, ANCOVA — [p-value comment as in outcome 1, analysis 1]; LS mean difference = 0.06, 95% CI 2-sided [0.02 to 0.11], Standard Error of Mean 0.022

3. Secondary Outcome: Change in Evening PEF From Baseline to the Treatment Period Average
Description: as for outcome 1
Time Frame: Baseline to 6 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: liters/minute
Arm/Group | Placebo | Budesonide
Number analyzed (Participants) | 150 | 151
liters/minute | 4.0 (3.08) | 14.7 (3.13)
Statistical Analysis 1: Comparison: Placebo vs Budesonide; Change from baseline to treatment period average was analyzed using an ANCOVA model with terms for treatment, age group (<8 years and ≥8 years of age) and country with baseline as a covariate; Test type: Superiority or Other; p = 0.0004, ANCOVA; LS mean difference = 10.8, 95% CI 2-sided [4.9 to 16.7], Standard Error of Mean 3.00

4. Secondary Outcome: Change in Forced Vital Capacity (FVC) From Baseline to Treatment Period Average
Description: FVC is the total volume of air expired after a full inspiration. Baseline was defined as the pre-dose assessment value measured at randomization (Visit 3), and the treatment period average was calculated as the mean of all available data recorded during the entire treatment period.
Time Frame: Baseline to 6 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | Placebo | Budesonide
Number analyzed (Participants) | 149 | 152
liters | 0.00 (0.021) | 0.04 (0.021)
Statistical Analysis 1: Comparison: Placebo vs Budesonide; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.0673, ANCOVA; LS mean difference = 0.04, 95% CI 2-sided [0.00 to 0.08], Standard Error of Mean 0.020

5. Secondary Outcome: Change in Forced Mid-expiratory Flow Between 25% and 75% of the FVC (FEF25-75) From Baseline to Treatment Period Average
Description: FEF25-75 is the average rate of airflow during the midportion of the forced vital capacity. Baseline was defined as the pre-dose assessment value measured at randomization (Visit 3), and the treatment period average was calculated as the mean of all available data recorded during the entire treatment period.
Time Frame: Baseline to 6 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: liters/second
Arm/Group | Placebo | Budesonide
Number analyzed (Participants) | 149 | 152
liters/second | 0.01 (0.045) | 0.11 (0.045)
Statistical Analysis 1: Comparison: Placebo vs Budesonide; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.0216, ANCOVA; LS mean difference = 0.10, 95% CI 2-sided [0.01 to 0.19], Standard Error of Mean 0.044

6. Secondary Outcome: Change in Total Daily and Daytime Asthma Symptom Scores From Baseline to Treatment Period Average
Description: Patients, with the help of their caregiver, were required to rate and document their asthma symptoms twice daily as an overall symptom score for the time period since their previous recording. The following rating scales were used: 0 = None; no symptoms of asthma; 1 = Mild symptoms; awareness of asthma symptoms and/or signs that are easily tolerated; 2 = Moderate symptoms, asthma symptoms with some discomfort, causing some interference with daily activities or sleep; 3 = Severe symptoms; incapacitating asthma symptoms and/or signs, with inability to perform daily activities or to sleep.
Time Frame: Baseline to 6 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Budesonide
Number analyzed (Participants) | 151 | 152
units on a scale
  Daytime asthma symptom score | -0.2 (0.06) | -0.4 (0.06)
  Total asthma symptom score | -0.5 (0.11) | -0.8 (0.11)
Statistical Analysis 1: Comparison: Placebo vs Budesonide; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.0004, ANCOVA — Analysis for change in daytime asthma symptom score from baseline to treatment period average; LS mean difference = -0.2, 95% CI 2-sided [-0.31 to -0.09], Standard Error of Mean 0.06
Statistical Analysis 2: Comparison: Placebo vs Budesonide; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.0015, ANCOVA — Analysis for change in total asthma symptom score from baseline to treatment period average; LS mean difference = -0.3, 95% CI 2-sided [-0.55 to -0.13], Standard Error of Mean 0.11

7. Secondary Outcome: Change in Nighttime Asthma Symptom Score From Baseline to Treatment Period Average
Description: as for outcome 6
Time Frame: Baseline to 6 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Budesonide
Number analyzed (Participants) | 152 | 152
units on a scale | -0.3 (0.06) | -0.4 (0.06)
Statistical Analysis 1: Comparison: Placebo vs Budesonide; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.0079, ANCOVA; LS mean difference = -0.1, 95% CI 2-sided [-0.26 to -0.04], Standard Error of Mean 0.06

8. Secondary Outcome: Change in Nighttime Awakenings and Nighttime Awakenings With Reliever Medication Use From Baseline to Treatment Period Average
Description: Patients, with the help of their caregiver, were asked to respond to a standard question each morning as they completed their eDiary. The question to be answered was, "Did your asthma cause you to wake-up last night?" If yes, patients were asked, "Did you need to use your reliever medication (albuterol/salbutamol inhaler) before you went back to sleep?" Baseline is defined as the percentage of days where patient experienced nighttime awakenings out of all available days where data was collected during the last 7 days of the run-in period.
Time Frame: Baseline to 6 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percentage of days with awakenings
Arm/Group | Placebo | Budesonide
Number analyzed (Participants) | 152 | 152
percentage of days with awakenings
  Nighttime awakenings | -9.8 (1.81) | -14.5 (1.84)
  Nighttime awakenings with reliever use | -6.1 (1.17) | -10.0 (1.18)
Statistical Analysis 1: Comparison: Placebo vs Budesonide; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.0095, ANCOVA — Analysis for change in nighttime awakenings from baseline to treatment period average; LS mean difference = -4.7, 95% CI 2-sided [-8.2 to -1.1], Standard Error of Mean 1.78
Statistical Analysis 2: Comparison: Placebo vs Budesonide; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.0007, ANCOVA — Analysis for change in nighttime awakenings with reliever medication use from baseline to treatment period average; LS mean difference = -3.9, 95% CI 2-sided [-6.2 to -1.7], Standard Error of Mean 1.15

9. Secondary Outcome: Change in Total Daily and Daytime Reliever Medication Use From Baseline to Treatment Period Average
Description: The patient, with the help of their caregiver, recorded the number of inhalations of reliever medication used, for relief of asthma symptoms, twice daily in the eDiary. Patients were asked to respond to a standard question twice daily (morning and evening). The question to be answered was, "How many albuterol/salbutamol inhalations since last diary entry?"
Time Frame: Baseline to 6 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: inhalations per day
Arm/Group | Placebo | Budesonide
Number analyzed (Participants) | 151 | 152
inhalations per day
  Daytime reliever medication use | -0.1 (0.07) | -0.4 (0.07)
  Total reliever medication use | -0.3 (0.11) | -0.7 (0.11)
Statistical Analysis 1: Comparison: Placebo vs Budesonide; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.0001, ANCOVA — Analysis for change in daytime reliever medication use from baseline to treatment period average; LS mean difference = -0.3, 95% CI 2-sided [-0.4 to -0.1], Standard Error of Mean 0.07
Statistical Analysis 2: Comparison: Placebo vs Budesonide; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA — Analysis for change in total reliever medication use from baseline to treatment period average; LS mean difference = -0.5, 95% CI 2-sided [-0.7 to -0.2], Standard Error of Mean 0.11

10. Secondary Outcome: Change in Nighttime Reliever Medication Use From Baseline to Treatment Period Average
Description: as for outcome 9
Time Frame: Baseline to 6 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: inhalations per day
Arm/Group | Placebo | Budesonide
Number analyzed (Participants) | 152 | 152
inhalations per day | -0.1 (0.06) | -0.4 (0.06)
Statistical Analysis 1: Comparison: Placebo vs Budesonide; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA; LS mean difference = -0.2, 95% CI 2-sided [-0.3 to -0.1], Standard Error of Mean 0.06

11. Secondary Outcome: Number of Withdrawals Due to Pre-defined Asthma Events
Description: Patients were considered to have experienced a "pre-defined asthma event" if any of the following conditions were met during the study: 1. At each visit or follow-up visit, a decrease in morning pre-dose FEV1 >=20% from the Visit 3 (randomization visit) morning pre-dose FEV1 or a decrease to <65% of predicted normal value; 2. The use of >=8 actuations of albuterol/salbutamol per day on 3 or more days within any period of 7 consecutive days following randomization; 3. A decrease in morning PEF >=20% from baseline on 3 or more days within any period of 7 consecutive days after randomization; 4. Two or more nights with an awakening due to asthma, which required the use of reliever medication within any period of 7 consecutive days after randomization; 5. A clinical exacerbation requiring emergency treatment, hospitalization, or use of an asthma medication not allowed by the study protocol.
Time Frame: Baseline to 6 weeks
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Placebo | Budesonide
Number analyzed (Participants) | 152 | 152
participants | 50 | 25
Statistical Analysis 1: Comparison: Placebo vs Budesonide; Test type: Superiority or Other; p = 0.0004, Log Rank

ADVERSE EVENTS:
Arm/Group | Budesonide pMDI 160mcg b.i.d. | Placebo pMDI b.i.d.
Serious Adverse Events (participants affected / at risk) | 0/152 | 0/152
Other Adverse Events (participants affected / at risk) | 27/152 | 40/152
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Budesonide pMDI 160mcg b.i.d. (N=152) | Placebo pMDI b.i.d. (N=152)
INFLUENZA (Infections and infestations) | 4 (5) | 4 (5)
NASOPHARYNGITIS (Infections and infestations) | 12 (12) | 9 (11)
PHARYNGITIS (Infections and infestations) | 5 (5) | 8 (8)
VIRAL UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 3 (3) | 8 (9)
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 11 (11)
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days